CLINICAL TRIAL: NCT01100307
Title: A Phase 3, Randomized, Controlled, Double-Masked, Multi-Center, Comparative, In Parallel Groups (For 24 Weeks), To Compare The Efficacy And Safety Of 0.3 MG Pegaptanib Sodium, With Sham Injections, And Open Study (For 30 Weeks) To Confirm The Safety Of 0.3 MG Pegaptanib Sodium In Subjects With Diabetic Macular Edema (DME)
Brief Title: A Phase 3 Study To Compare The Efficacy And Safety Of 0.3 MG Pegaptanib Sodium To Sham Injections In Subjects With Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5751034
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-05

CONDITIONS: Macular Edema; Diabetic Mellitus; Retinal Disease
Keywords: diabetic macular edema; Macugen; sham-controlled study
MeSH Terms: conditions — Macular Edema; Retinal Diseases | interventions — pegaptanib; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pegaptanib sodium (Experimental)
  Interventions: Drug: pegaptanib sodium
- sham injection (Sham Comparator)
  Interventions: Other: sham injection

INTERVENTIONS:
Drug: pegaptanib sodium — Intravitreal injection of 0.3 mg every 6 weeks
  Arms: pegaptanib sodium
Other: sham injection — sham injection every 6 weeks
  Arms: sham injection

SUMMARY:
The purpose of the study to assess the efficacy of pegaptanib sodium 0.3 mg comparing sham injection and to confirm safety of pegaptanib sodium 0.3 mg in subjects with diabetic macular edema.

DETAILED DESCRIPTION:
During the study, an issue was reported concerning proper maintenance of treatment masking (See Result: Limitations and Caveats)

ELIGIBILITY:
Inclusion Criteria:

* Type I, or Type II diabetic subjects
* Subjects must have macular edema that involves the center field of the macula 3. Foveal thickness of at least 250 μm 4. Best corrected distance visual acuity in the study eye must be a letter score between 68 and 35 inclusive

Exclusion Criteria:

* Eyes with prior panretinal photocoagulation (PRP) less than 4 months prior to baseline eyes in which PRP is needed now or is likely to be needed within the next 9 months
* HbA1C level >12% or recent signs of uncontrolled diabetes
* Atrophy/scarring/fibrosis involving the center of the macula, including evidence of laser treated atrophy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- Japan (43):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - Aomori Prefectural Chuo Hospital, Aomori, Aomori
  - Chiba University Hospital, Chiba, Chiba
  - Juntendo University Hospital Urayasu, Ophthalmology, Urayasu-shi, Chiba
  - Hayashi Eye Hospital, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Murakami Karindo Hospital, Fukuoka, Fukuoka
  - Ohshima Hospital of Ophthalmology, Fukuoka, Fukuoka
  - St. Mary's Hospital, Kurume, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gunma University Hospital, Maebashi, Gunma
  - Kimura Eye & Internal Medicine Hospital, Kure, Hiroshima
  - Asahikawa Medical College Hospital, Asahikawa, Hokkaido
  - Yoshida Eye Hospital, Hakodate, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Amagasaki Hospital, Amagasaki, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kohnan Hospital, Kobe, Hyōgo
  - Hitachi General Hospital, Hitachi, Ibaraki
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Kagawa University Hospital, Kida-gun, Kagawa-ken
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Ideta eye hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - NTT East Tohoku Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto, Nagano
  - Nara Medical University Hospital, Kashihara, Nara
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Osaka City University Hospital, Osaka, Osaka
  - Osaka general medical center, Osaka, Osaka
  - Osaka Saiseikai Izou Hospital, Osaka, Osaka
  - Kinki University Hospital, Anesthesiology, Osaka-sayama-shi, Osaka
  - Saga Prefectural Hospital Koseikan, Saga, Saga-ken
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Nihon University Surugadai Hospital, Chiyoda-ku, Tokyo
  - Ochanomizu Inoue Eye Clinic, Chiyoda-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Hirota Eye Clinic, Shūnan, Yamaguchi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751034&StudyName=A%20Phase%203%20Study%20To%20Compare%20The%20Efficacy%20And%20Safety%20Of%200.3%20MG%20Pegaptanib%20Sodium%20To%20Sham%20Injections%20In%20Subjects%20With%20Diabetic%20Macula

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegaptanib Sodium: Pegaptanib sodium 0.3 milligrams were administered as an intravitreous injection every 6 weeks. Total number of injections were 4 times in the double masked phase (up to Week 24) and 5 times in the open phase (from Week 24 to Week 54).
- Sham in Double Masked, Then Pegaptanib Sodium in Open Phase: Sham injection was conducted during the double masked phase (up to Week 24) according to the identical procedure of pegaptanib sodium administration, with exceptions of no needle used and no medication. Pegaptanib sodium 0.3 milligrams were administered as an intravitreous injection every 6 weeks in participants who were originally randomized to Sham and entered in the open phase (Week 24 to Week 54). Total number of injection was 5 times in the open phase.
Period: Double Masked Phase (Up to Week 24)
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Started | 123 | 120
Completed | 117 | 116
Not Completed | 6 | 4
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 5 | 2
Period: Open Phase (Week 24 up to Week 54)
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Started | 116 (One participant discontinued from the study due to adverse event before study drug administration.) | 112 (Four participants did not enter to the open phase after completing the double masked phase.)
Completed | 110 | 99
Not Completed | 6 | 13
Not completed — Lack of Efficacy | 1 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase | Total
Number analyzed (Participants) | 123 | 120 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 49 | 101
  >=65 years | 71 | 71 | 142
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 55 | 113
  Male | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience a ≥10 Letter Improvement of Visual Acuity (VA) in Early Treatment Diabetic Retinopathy Study (ETDRS) Chart From Baseline at Week 24: Double Masked Phase
Description: Best-corrected visual acuity (VA) measurements were performed using retro-illuminated, modified Ferris-Bailey Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Time Frame: Baseline and Week 24
Population: Full Analysis Set 1: participants who received at least 1 injection after randomized to study treatment and had VA assessments both at baseline and at least once at post-dose in the double-masked phase. Missing values except for baseline value were imputed using a last observation carried forward approach (LOCF).
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 123 | 120
Participants | 25 | 6
Statistical Analysis 1: Comparison: Pegaptanib Sodium vs Sham in Double Masked, Then Pegaptanib Sodium in Open Phase; The null hypothesis was to assume that there was no difference between the pegaptanib sodium and sham injection groups. The alternative was to assume that there was difference between the pegaptanib sodium and sham injection groups; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel — Significance level of test in the comparison between pegaptanib sodium 0.3 mg and sham was set to 0.05; Stratification factors (HbA1c and baseline visual acuity categories); Odds Ratio (OR) = 4.85, 95% CI 2-sided [1.92 to 12.28]

2. Secondary Outcome: Change From Baseline in Visual Acuity (VA): Double Masked Phase
Description: Changes in VA were monitored through refraction and best-corrected VA measurements using retro-illuminated, modified Ferris-Bailey ETDRS charts
Time Frame: Baseline, Weeks 6, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 123 | 120
Letters
  Week 6 | 2.7 (5.39) | 0.2 (5.90)
  Week 12 | 3.2 (6.19) | -0.6 (8.60)
  Week 18 | 2.8 (7.84) | 0.1 (8.14)
  Week 24 | 3.1 (7.50) | -1.2 (8.80)
Statistical Analysis 1: Comparison: Pegaptanib Sodium vs Sham in Double Masked, Then Pegaptanib Sodium in Open Phase; Comparison at Week 6: The null hypothesis was to assume that there was no difference between the pegaptanib sodium and sham injection groups. The alternative was to assume that there was difference between the pegaptanib sodium and sham injection groups; Test type: Superiority or Other; p = 0.0006, ANCOVA — Significance level of test in the comparison between pegaptanib sodium 0.3 mg and sham was set to 0.05; Based on an analysis of covariance with treatment as a factor and stratification factors (HbA1c and baseline visual acuity categories) as covariates; Mean Difference (Final Values) = 2.52, 95% CI 2-sided [1.10 to 3.94]
Statistical Analysis 2: Comparison: Pegaptanib Sodium vs Sham in Double Masked, Then Pegaptanib Sodium in Open Phase; Comparison at Week 12: The null hypothesis was to assume that there was no difference between the pegaptanib sodium and sham injection groups. The alternative was to assume that there was difference between the pegaptanib sodium and sham injection groups; Test type: Superiority or Other; p = 0.0001, ANCOVA — Significance level of test in the comparison between pegaptanib sodium 0.3 mg and sham was set to 0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 3.69, 95% CI 2-sided [1.81 to 5.58]
Statistical Analysis 3: Comparison: Pegaptanib Sodium vs Sham in Double Masked, Then Pegaptanib Sodium in Open Phase; Comparison at Week 18: The null hypothesis was to assume that there was no difference between the pegaptanib sodium and sham injection groups. The alternative was to assume that there was difference between the pegaptanib sodium and sham injection groups; Test type: Superiority or Other; p = 0.0096, ANCOVA — Significance level of test in the comparison between pegaptanib sodium 0.3 mg and sham was set to 0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.65, 95% CI 2-sided [0.65 to 4.65]
Statistical Analysis 4: Comparison: Pegaptanib Sodium vs Sham in Double Masked, Then Pegaptanib Sodium in Open Phase; Comparison at Week 24: The null hypothesis was to assume that there was no difference between the pegaptanib sodium and sham injection groups. The alternative was to assume that there was difference between the pegaptanib sodium and sham injection groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level of test in the comparison between pegaptanib sodium 0.3 mg and sham was set to 0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 4.26, 95% CI 2-sided [2.19 to 6.32]

3. Secondary Outcome: Number of Participants Underwent Focal/Grid Laser, or Vitrectomy: Double Masked Phase
Description: Included focal laser photocoagulation, grid laser photocoagulation, and vitrectomy.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 123 | 120
Participants
  Focal/Grid Lase | 3 | 1
  Vitrectomy | 0 | 1

4. Secondary Outcome: Number of Participants Who Experience a ≥10 Letter Improvement of Visual Acuity in Early Treatment Diabetic Retinopathy Study (ETDRS) Chart From Baseline at Week 54: Open Phase
Description: as for outcome 1
Time Frame: Baseline and Week 54
Population: Full Analysis Set 2: participants who received at least 1 injection and had VA assessments both at baseline and at least once at post-dose in open phase. Missing values except for baseline value were imputed using a last observation carried forward approach (LOCF).
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 116 | 112
Participants | 28 | 15

5. Secondary Outcome: Change From Baseline in Visual Acuity (VA): Open Phase
Description: Changes in VA were monitored through refraction and best-corrected VA measurements using retro-illuminated, modified Ferris-Bailey Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Time Frame: Baseline, Weeks 30, 36, 42, 48 and 54
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 116 | 112
Letters
  Week 30 | 3.5 (8.62) | -0.1 (7.78)
  Week 36 | 4.4 (8.43) | 0.6 (7.91)
  Week 42 | 4.3 (8.27) | 0.3 (8.86)
  Week 48 | 4.1 (8.52) | -0.8 (10.09)
  Week 54 | 3.6 (8.93) | -0.5 (10.48)

6. Secondary Outcome: Number of Participants Who Underwent Focal/Grid Laser, or Vitrectomy: Open Phase
Description: Included focal laser photocoagulation, grid laser photocoagulation, and vitrectomy.
Time Frame: Weeks 24 to 54
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 116 | 112
Participants
  Focal/Grid Laser | 3 | 3
  Vitrectomy | 0 | 0

7. Other Pre Specified Outcome: Mean Visual Acuity Over Time at Each Time Point: Double Masked Phase
Description: as for outcome 1
Time Frame: Baseline, Weeks 6, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 123 | 120
Letters
  Baseline | 56.8 (8.39) | 56.9 (8.15)
  Week 6 | 59.5 (8.24) | 57.1 (10.29)
  Week 12 | 60.0 (9.32) | 56.4 (11.65)
  Week 18 | 59.7 (9.66) | 57.1 (11.52)
  Week 24 | 59.9 (9.89) | 55.7 (12.18)

8. Other Pre Specified Outcome: Distribution of Change From Baseline of Visual Acuity (VA) at Each Time Point: Double Masked Phase
Description: Best-corrected VA measurements were performed using retro-illuminated, modified Ferris-Bailey ETDRS charts.
  Change from baseline in VA was categorized as follows: Lost 15 letters or more; Lost 10 - 14 letters; Lost 1 - 9 Letters; No change or gained 1 - 9 letters; Gained 10 - 14 letters; Gained 15 letters or more.
Time Frame: Baseline, Weeks 6, 12, 18, and 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 123 | 120
Participants
  Week 6: Lost 15 Letters or More | 1 | 4
  Week 6: Lost 10 - 14 Letters | 0 | 2
  Week 6: Lost 1 - 9 Letters | 33 | 40
  Week 6: No Change/Gained 1 - 9 Letters | 74 | 71
  Week 6: Gained 10 - 14 Letters | 12 | 3
  Week 6: Gained 15 Letters or More | 3 | 0
  Week 12: Lost 15 Letters or More | 1 | 5
  Week 12: Lost 10 - 14 Letters | 1 | 3
  Week 12: Lost 1 - 9 Letters | 28 | 50
  Week 12: No Change/Gained 1 - 9 Letters | 76 | 54
  Week 12: Gained 10 - 14 Letters | 12 | 7
  Week 12: Gained 15 Letters or More | 5 | 1
  Week 18: Lost 15 Letters or More | 2 | 4
  Week 18: Lost 10 - 14 Letters | 3 | 3
  Week 18: Lost 1 - 9 Letters | 33 | 43
  Week 18: No Change/Gained 1 - 9 Letters | 61 | 62
  Week 18: Gained 10 - 14 Letters | 15 | 6
  Week 18: Gained 15 Letters or More | 9 | 2
  Week 24: Lost 15 Letters or More | 1 | 9
  Week 24: Lost 10 - 14 Letters | 6 | 5
  Week 24: Lost 1 - 9 Letters | 30 | 41
  Week 24: No Change/Gained 1 - 9 Letters | 61 | 59
  Week 24: Gained 10 - 14 Letters | 18 | 5
  Week 24: Gained 15 Letters or More | 7 | 1

9. Other Pre Specified Outcome: Number of Participants Who Experience a ≥10 Letter Improvement of Visual Acuity in Early Treatment Diabetic Retinopathy Study (ETDRS) Chart From Baseline: Double Masked Phase
Description: as for outcome 1
Time Frame: Baseline, Weeks 6, 12, 18, and 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 123 | 120
Participants
  Week 6 | 15 | 3
  Week 12 | 17 | 8
  Week 18 | 24 | 8
  Week 24 | 25 | 6

10. Other Pre Specified Outcome: Number of Participants Who Experience a ≥15, ≥5, or ≥0 Letter Improvement of Visual Acuity in Early Treatment Diabetic Retinopathy Study (ETDRS) Chart From Baseline at Week 24: Double Masked Phase
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 123 | 120
Participants
  ≥15 Letter Improvement | 7 | 1
  ≥5 Letter Improvement | 49 | 31
  ≥0 Letter Improvement | 86 | 65

11. Other Pre Specified Outcome: Number of Participants Exhibiting a Decrease From Baseline in Retinal Thickness at the Center Point by ≥25 Percent and ≥50 Percent Using Optical Coherence Tomography (OCT) at Week 24: Double Masked Phase
Description: OCT, a noninvasive, noncontact, transpupillary imaging technology, was utilized to image retinal structures in vivo. The anatomic layers within the retina, retinal thickness could be measured.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 123 | 120
Participants
  ≥25% Decrease From Baseline | 42 | 25
  ≥50% Decrease From Baseline | 11 | 8

12. Other Pre Specified Outcome: Change From Baseline in National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) Composite Score/Sub-scale Score at Week 24: Double Masked Phase
Description: NEI-VFQ 25, Japanese version v.1.4 for self-administering questionnaires consisted of the base set of 25 questions and 12 subscale scores.
  Response categories to each question were converted to a 0 to 100 scale so that the lowest and highest possible scores were set at 0 and 100 points, respectively. A higher score represented better functioning. Questions within each sub-scale were averaged together to create the 12 sub-scale scores. The overall composite score was calculated by averaging the vision-targeted subscale scores excluding the general health-rating question.
  Positive change indicated improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 123 | 120
Units on a scale
  General Health (n=123, 118) | -0.2 (18.80) | -2.1 (20.56)
  General Vision (n=123, 118) | 2.8 (17.80) | 0.7 (19.20)
  Ocular Pain (n=123, 118) | -0.5 (18.35) | 0.6 (18.77)
  Near Vision Activities (n=123, 118) | -0.5 (19.01) | 0.6 (18.60)
  Distance Vision Activities (n=123, 118) | 0.5 (15.92) | -1.3 (15.80)
  Social Functioning (n=123, 117) | 0.7 (17.77) | -1.7 (17.13)
  Mental Health (n=123, 118) | 0.5 (19.05) | -0.5 (17.91)
  Role Difficulties (n=123, 118) | -1.6 (23.36) | -1.1 (21.72)
  Dependency (n=123, 118) | -0.1 (18.11) | -1.1 (18.38)
  Driving (n=80, 73) | -1.4 (14.34) | -5.7 (20.84)
  Color Vision (n=119, 115) | 2.9 (15.67) | -0.9 (19.85)
  Peripheral Vision (n=123, 117) | 1.4 (23.15) | -4.1 (21.26)
  Composite Score (n=123, 118) | 0.5 (10.37) | -1.1 (10.85)

13. Other Pre Specified Outcome: Mean Visual Acuity Over Time at Each Time Point: Open Phase
Description: as for outcome 1
Time Frame: Baseline, Weeks 30, 36, 42, 48, and 54
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 116 | 112
Letters
  Baseline | 57.2 (8.07) | 56.7 (8.28)
  Week 30 | 60.7 (10.52) | 56.6 (11.25)
  Week 36 | 61.6 (10.47) | 57.3 (11.59)
  Week 42 | 61.5 (10.01) | 57.0 (12.24)
  Week 48 | 61.3 (10.11) | 55.9 (13.61)
  Week 54 | 60.8 (10.63) | 56.2 (13.71)

14. Other Pre Specified Outcome: Distribution of Change From Baseline of Visual Acuity (VA) at Each Time Point: Open Phase
Description: as for outcome 8
Time Frame: Baseline, Weeks 30, 36, 42, 48, and 54
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 116 | 112
Participants
  Week 30: Lost 15 Letters or More | 4 | 8
  Week 30: Lost 10 - 14 Letters | 2 | 5
  Week 30: Lost 1 - 9 Letters | 31 | 31
  Week 30: No Change or Gained 1 - 9 Letters | 53 | 61
  Week 30: Gained 10 - 14 Letters | 15 | 7
  Week 30: Gained 15 Letters or More | 11 | 0
  Week 36: Lost 15 Letters or More | 3 | 6
  Week 36: Lost 10 - 14 Letters | 1 | 8
  Week 36: Lost 1 - 9 Letters | 22 | 25
  Week 36: No Change or Gained 1 - 9 Letters | 64 | 63
  Week 36: Gained 10 - 14 Letters | 13 | 10
  Week 36: Gained 15 Letters or More | 13 | 0
  Week 42: Lost 15 Letters or More | 2 | 8
  Week 42: Lost 10 - 14 Letters | 2 | 10
  Week 42: Lost 1 - 9 Letters | 24 | 26
  Week 42: No Change or Gained 1 - 9 Letters | 59 | 53
  Week 42: Gained 10 - 14 Letters | 16 | 12
  Week 42: Gained 15 Letters or More | 13 | 3
  Week 48: Lost 15 Letters or More | 2 | 13
  Week 48: Lost 10 - 14 Letters | 5 | 9
  Week 48: Lost 1 - 9 Letters | 27 | 24
  Week 48: No Change or Gained 1 - 9 letters | 51 | 54
  Week 48: Gained 10 - 14 Letters | 15 | 9
  Week 48: Gained 15 Letters or More | 16 | 3
  Week 54: Lost 15 Letters or More | 3 | 10
  Week 54: Lost 10 - 14 Letters | 3 | 10
  Week 54: Lost 1 - 9 Letters | 27 | 28
  Week 54: No Change or Gained 1 - 9 Letters | 55 | 49
  Week 54: Gained 10 - 14 Letters | 15 | 13
  Week 54: Gained 15 Letters or More | 13 | 2

15. Other Pre Specified Outcome: Number of Participants Who Experience a ≥10 Letter Improvement of Visual Acuity in Early Treatment Diabetic Retinopathy Study (ETDRS) Chart From Baseline: Open Phase
Description: as for outcome 1
Time Frame: Baseline, Weeks 30, 36, 42, 48, and 54
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 116 | 112
Participants
  Week 30 | 26 | 7
  Week 36 | 26 | 10
  Week 42 | 29 | 15
  Week 48 | 31 | 12
  Week 54 | 28 | 15

16. Other Pre Specified Outcome: Number of Participants Who Experience a ≥15, ≥5, or ≥0 Letter Improvement of Visual Acuity in Early Treatment Diabetic Retinopathy Study (ETDRS) Chart From Baseline at Week 54: Open Phase
Description: as for outcome 1
Time Frame: Baseline and Week 54
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 116 | 112
Participants
  ≥15 Letter Improvement | 13 | 2
  ≥5 Letter Improvement | 45 | 40
  ≥0 Letter Improvement | 83 | 64

17. Other Pre Specified Outcome: Number of Participants Exhibiting a Decrease From Baseline in Retinal Thickness at the Center Point by ≥25 Percent and ≥50 Percent Using Optical Coherence Tomography (OCT) at Week 54: Open Phase
Description: Retinal thickness was assessed by spectral-domain optical coherence tomography or OCT3000, a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
Time Frame: Baseline and Week 54
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 116 | 112
Participants
  ≥25% Decrease From Baseline | 56 | 38
  ≥50% Decrease From Baseline | 21 | 16

18. Other Pre Specified Outcome: Change From Baseline in The 25-Item National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) Composite Score/Sub-scale Score at Week 54: Open Phase
Description: as for outcome 12
Time Frame: Baseline and Week 54
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pegaptanib Sodium | Sham in Double Masked, Then Pegaptanib Sodium in Open Phase
Number analyzed (Participants) | 116 | 112
Units on a scale
  General Health (n=116, 110) | -1.5 (20.13) | -1.8 (20.52)
  General Vision (n=116, 110) | 4.7 (15.68) | 0.7 (17.96)
  Ocular Pain (n=116, 110) | 1.8 (17.15) | 0.0 (17.35)
  Near Vision Activities (n=116, 110) | 1.5 (17.28) | -0.6 (19.92)
  Distance Vision Activities (n=116, 110) | 1.4 (15.97) | -0.5 (15.46)
  Social Functioning (n=116, 110) | -2.5 (17.92) | -2.5 (17.25)
  Mental Health (n=116, 110) | 2.1 (19.85) | -2.7 (20.43)
  Role Difficulties (n=116, 110) | 0.5 (23.34) | -0.6 (20.90)
  Dependency (n=116, 110) | 0.9 (19.30) | -3.3 (18.76)
  Driving (n=74, 69) | -2.0 (18.28) | -7.2 (26.03)
  Color Vision (n=112, 109) | -0.4 (15.00) | -2.8 (18.43)
  Peripheral Vision (n=115, 110) | 0.9 (22.20) | -3.4 (22.07)
  Composite Score (n=116, 110) | 0.8 (11.15) | -1.8 (11.16)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Pegaptanib Sodium (Baseline to Week 24): Pegaptanib sodium 0.3 milligrams were administered as an intravitreous injection every 6 weeks. Total number of injections were 4 times in the double masked phase (up to Week 24).
- Sham (Baseline to Week 24): Sham injection was conducted during the double masked phase (up to Week 24) according to the identical procedure of pegaptanib sodium administration, with exceptions of no needle used and no medication.
- Pegaptanib Sodium (Baseline to Week 54): Pegaptanib sodium 0.3 milligrams were administered as an intravitreous injection every 6 weeks. Total number of injections were 4 times in the double masked phase (up to Week 24) and 5 times in the open phase (from Week 24 to Week 54).
- Sham Conversion (Week 24 to Week 54): Pegaptanib sodium 0.3 milligrams were administered as an intravitreous injection every 6 weeks in participants who were originally randomized to Sham and entered in the open phase (Week 24 to Week 54). Total number of injection was 5 times in the open phase.
Arm/Group | Pegaptanib Sodium (Baseline to Week 24) | Sham (Baseline to Week 24) | Pegaptanib Sodium (Baseline to Week 54) | Sham Conversion (Week 24 to Week 54)
Serious Adverse Events (participants affected / at risk) | 10/123 | 10/120 | 19/123 | 7/112
Other Adverse Events (participants affected / at risk) | 72/123 | 53/120 | 83/123 | 40/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegaptanib Sodium (Baseline to Week 24) (N=123) | Sham (Baseline to Week 24) (N=120) | Pegaptanib Sodium (Baseline to Week 54) (N=123) | Sham Conversion (Week 24 to Week 54) (N=112)
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 1 | 1
Diabetic retinal oedema (Eye disorders) | 0 | 3 | 1 | 1
Glaucoma (Eye disorders) | 2 | 0 | 2 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Viral myositis (Infections and infestations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 1 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Rhabdomyclysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegaptanib Sodium (Baseline to Week 24) (N=123) | Sham (Baseline to Week 24) (N=120) | Pegaptanib Sodium (Baseline to Week 54) (N=123) | Sham Conversion (Week 24 to Week 54) (N=112)
Conjunctival Haemorrhage (Eye disorders) | 54 | 33 | 57 | 4
Conjunctival Oedema (Eye disorders) | 12 | 13 | 12 | 0
Corneal Erosion (Eye disorders) | 3 | 5 | 8 | 2
Diabetic Retinal Oedema (Eye disorders) | 7 | 4 | 13 | 11
Eye pain (Eye disorders) | 9 | 1 | 11 | 1
Punctate Keratitis (Eye disorders) | 12 | 7 | 17 | 7
Nasopharyngitis (Infections and infestations) | 15 | 11 | 27 | 10
Intraocular Pressure Increased (Investigations) | 8 | 0 | 18 | 10
Conjunctival hyperaemia (Eye disorders) | 2 | 7 | 2 | 0

LIMITATIONS AND CAVEATS:
During the study, an issue was reported concerning proper maintenance of treatment masking. Due to this masking process issue, the study results cannot be interpreted as that arising from a well-controlled double-masked trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.